CLINICAL TRIAL: NCT02836457
Title: ELIQUIS (APIXABAN) Regulatory Post-Marketing Surveillance In Clinical Practice for Venous Thromboembolism (VTE) Treatment and Prevention Of Recurrent VTE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-396
Record Dates: First submitted 2016-07-12; First posted 2016-07-19 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Population with Exposure to ELIQUIS (APIXABAN)

SUMMARY:
The primary objectives of this study is to estimate the real-world safety profile of Eliquis in Japanese Venous Thromboembolism patients and to estimate the risk factors likely to affect the incidence of bleeding. Lastly, the secondary objective of this study is to estimate the real-world effectiveness profile of Eliquis in Japanese Venous Thromboembolism patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are initiating Eliquis for the treatment of VTE or prevention of recurrent VTE for the first time

Exclusion Criteria:

* Prior treatment with Eliquis for nonvalvular atrial fibrillation or VTE
* Patients initiating Eliquis for the treatment of atrial fibrillation
* Off-label use of Eliquis

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 1134 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence of all treatment-related adverse events ( AE) | 52 Weeks
The incidence of serious adverse events (SAE) | 52 Weeks
The incidence of unexpected treatment-related adverse events | 52 Weeks
  The incidence of unexpected treatment-related adverse events will be analyzed by seriousness, causality, and outcomes of adverse events
The incidence of bleeding | 52 Weeks
  The incidence of bleeding will be analyzed by seriousness, causality, and outcomes of adverse events

SECONDARY OUTCOMES:
The incidence of venous thromboembolism (VTE) | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html